CLINICAL TRIAL: NCT02256072
Title: Advance Planning for Home Services for Seniors
Acronym: APHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lee Lindquist, Associate Professor of Medicine, Associate Division Chief of Geriatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IH-12-11-4259
Record Dates: First submitted 2014-09-25; First posted 2014-10-03 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Alzheimers, Falls, Aging in Place
Keywords: aging, geriatrics, aging in place, home services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plan Your Lifespan Website (Experimental): Participants in the intervention arm will navigate the Plan Your Lifespan website, a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. The Plan Your Lifespan tool is also interactive in that it allows participants to enter their information and share it with others to facilitate conversations and decision-making.
  Interventions: Other: Plan Your Lifespan Website
- Go4Life Website (Other): Participants in the attention control arm will navigate an electronic educational session via a National Institute on Aging at NIH Website, Go4Life, a website about physical activity and exercise as it is a topic of interest to seniors. Our attention control group will control for the possibility that regular contact with the study team may improve outcomes in participants randomized to the intervention website.
  Interventions: Other: Go4Life Website

INTERVENTIONS:
Other: Plan Your Lifespan Website — Participants in the intervention arm will navigate the advance planning tool, Plan Your Lifespan, a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. A minimum of 15 minutes and a maximum of 45 minutes will be allotted for navigating this website.The Plan Your Lifespan website is also interactive in that it allows participants to enter their information and share it with others to facilitate conversations and decision-making.
  Arms: Plan Your Lifespan Website
Other: Go4Life Website — Participants in the attention control arm will navigate an electronic educational session via a National Institute on Aging at NIH Website, Go4Life, a website about physical activity and exercise as it is a topic of interest to seniors. A minimum of 15 minutes and a maximum of 45 minutes will be allotted for navigating the website. The website is interactive and comparable to the intervention tool: http://go4life.nia.nih.gov/get-started).
  Other Names: National Institute on Aging at NIH Website
  Arms: Go4Life Website

SUMMARY:
The goal of this study is to develop and test an advance planning tool to help seniors understand projected health needs and plan ways to remain in their own homes when these crises occur. In this phase of the study through partnerships with seniors, senior community groups, area agencies on aging, and home care agencies the investigators are conducting a two-armed (attention control and intervention) randomized controlled trial.

Individuals will be randomly assigned to one of two interventions: attention control or the advance planning tool. The investigators attention control group will control for the possibility that regular contact with the study team may improve outcomes in participants randomized to the intervention website. Participants in the attention control arm will navigate an electronic educational session via a National Institute on Aging at NIH Web site about physical activity and exercise as it is a topic of interest to seniors. A minimum of 15 minutes and a maximum of 45 minutes will be allotted for navigating the Web site. The Web site is interactive and comparable to the intervention tool: http://go4life.nia.nih.gov/get-started).

If randomized to intervention, subjects will be introduced to the advance planning tool, the Plan Your Lifespan website, and given instructions on how to use it. Plan Your Lifespan is a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. The Plan Your Lifespan website is also interactive in that it allows participants to enter their information and share it with others to facilitate conversations and decision-making. Participants will navigate and complete the Web-based advance planning tool and will be allotted a minimum of 15 minutes and a maximum of 45 minutes to navigate the tool as part of the study.

All participants will be administered a pre- and post-test before and after viewing the website they were randomized to. All participants will be followed up at one and three months post via a brief phone call where follow-up questions will be asked of all participants.

DETAILED DESCRIPTION:
Seniors over the age of 65 years represent 13.1% of the United States population, with a projected 36% increase to 55 million by the year 2020. With advancing age, seniors experience an increased prevalence in memory loss, physical disability, and multiple chronic conditions (e.g., heart disease, emphysema, stroke, diabetes, cancers, hypertension, arthritis, osteoporosis, and macular degeneration). A large fear among seniors is loss of independence and removal from their homes to be placed in a nursing home. Seniors who remain in their own homes tend to have greater satisfaction, less depression, and maintain their physical function better than seniors residing in assisted living or nursing homes. Although remaining in the home is of utmost importance, many frail seniors teeter between safe living and personal endangerment. Falls, illness, and worsening memory all jeopardize a senior's independence and ability to remain in his or her home.

The advance planning tool, Plan Your Lifespan, provides information that will help older Americans to "fill in the gaps" in their lives as necessary. An established plan would offer guidance toward obtaining those resources and professional services that would be useful to the senior. An effective plan would be dynamic and adaptable to the senior's changing health needs.

The aim of this study is to conduct a randomized controlled trial of the advance planning tool to determine subject understanding of home care services, advanced health planning, and other patient-centered outcomes. The investigators also hypothesize the following:

H1: Compared to participants in the attention control group and controlling for baseline assessments, participants receiving the advance planning tool will show increased planning with regard to implementation/behavior, perception, and intention (measured via the Planning Assessment tool) one month after intervention.

H2: Compared to participants in the attention control group and controlling for baseline assessments, participants receiving the advance planning tool will show increased confidence in accessing home services (measured via the Confidence in Accessing Home Services tool) one month after intervention.

H3: Compared to participants in the attention control group and controlling for baseline assessments, participants receiving the advance planning tool will show increased understanding of home services (measured via the Understanding of Home Services tool) one month after intervention.

H4: Compared to participants in the attention control group and controlling for baseline assessments, participants receiving the advance planning tool will be more likely to report communicating their preferences about issues related to lifespan planning to people who may need to make decisions for them (measured via the Communication about Lifespan Planning Questionnaire) after study intervention.

H5: Compared to participants in the attention control group, participants randomized to the advance planning tool will report overall satisfaction with the intervention/attention control (measured via the Satisfaction with Intervention tool).

The total duration of the intervention for each participant will be three months with assessments at baseline, post-intervention, and two follow-up assessments at one and three months for a total of 4 data collection points.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* English speaking
* Score ≥ 4 questions correctly on the Brief Cognitive screener
* Self-identified comfort using a computer
* Self-identified comfort using the Internet to navigate a Website
* Have not previously participated in study's focus groups or pilot study

Exclusion Criteria:

* Less than age 65
* Non-English speaking
* Score < 4 questions correctly on the Brief Cognitive screener
* Not comfortable using a computer
* Not comfortable using the Internet to navigate a Website
* Previous participation in this study's focus groups or pilot study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 385 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee A Lindquist, MD, MPH, MBA, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Aging & In-Home Services of Northeast Indiana, Fort Wayne, Indiana

REFERENCES:
- [Derived] Lindquist LA, Ramirez-Zohfeld V, Sunkara PD, Forcucci C, Campbell DS, Mitzen P, Ciolino JD, Kricke G, Seltzer A, Ramirez AV, Cameron KA. Helping Seniors Plan for Posthospital Discharge Needs Before a Hospitalization Occurs: Results from the Randomized Control Trial of PlanYourLifespan.org. J Hosp Med. 2017 Nov;12(11):911-917. doi: 10.12788/jhm.2798. Epub 2017 Aug 23. PMID 29091979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study took place between October 1, 2014 and September 30, 2015.
Pre-assignment Details: Enrolled participants were excluded from the trial before assignment to groups if they did not reach randomization (e.g. they did not reach ). All participants reached randomization.
Groups:
- Plan Your Lifespan Website: Participants in the intervention arm will navigate PlanYourLifespan.org.
Period: Overall Study
Arm/Group | Plan Your Lifespan Website | Go4Life Website
Started | 194 | 191
Completed 1 Month Follow-Up | 167 (Completed the 1-month follow-up) | 179
Completed | 152 (Completed the 3-month follow-up) | 162
Not Completed | 42 | 29

BASELINE CHARACTERISTICS:
Groups:
- Plan Your Lifespan Website: Participants in the intervention arm will navigate Planyourlifespan.org, a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. The Plan Your Lifespan tool is also interactive in that it allows participants to enter their information and share it with others to facilitate conversations and decision-making.
  Plan Your Lifespan Website: Participants in the intervention arm will navigate the advance planning tool, Plan Your Lifespan, a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. A minimum of 15 minutes and a maximum of 45 minutes will be allotted for navigating this website.The Plan Your Lifespan website is also inte
- Total: Total of all reporting groups
Arm/Group | Plan Your Lifespan Website | Go4Life Website | Total
Number analyzed (Participants) | 194 | 191 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.67 (5.56) | 72.05 (5.57) | 71.86 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 157 | 306
  Male | 45 | 34 | 79
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 117 | 125 | 242
  Black or African American | 55 | 38 | 93
  Hispanic | 8 | 9 | 17
  Other | 5 | 5 | 10
  More than one race | 9 | 14 | 23
Marital Status [Number; unit: participants]
  Single, never married | 23 | 27 | 50
  Married | 85 | 75 | 160
  Widowed | 36 | 44 | 80
  Divorced/Separated | 50 | 45 | 95
Education [Number; unit: participants] — Reported education
  participants
    High school or less | 40 | 33 | 73
    Some college | 59 | 55 | 114
    College graduate | 95 | 103 | 198
Household Income [Number; unit: participants] — Self-reported combined annual household income.
  participants
    less than $20,000 | 43 | 45 | 88
    $20,000-$40,000 | 54 | 50 | 104
    $40,001-$60,000 | 27 | 31 | 58
    $60,001-$80,000 | 26 | 25 | 51
    $80,001-$100,000 | 17 | 19 | 36
    More than $100,000 | 18 | 13 | 31
    Not Sure/Don't Know | 2 | 4 | 6
    Prefer not to say | 7 | 4 | 11
Self-Reported Health Rating [Number; unit: participants]
  Poor | 4 | 4 | 8
  Fair | 18 | 22 | 40
  Good | 81 | 76 | 157
  Very Good | 70 | 62 | 132
  Excellent | 21 | 27 | 48
Living Arrangement [Number; unit: participants] — Self-reported current living arrangement.
  participants
    Live alone | 94 | 104 | 198
    Live with one other person | 90 | 75 | 165
    Live with multiple people (more than one) | 10 | 12 | 22
REALM-R [Number; unit: participants] — REALM-R score.
  participants
    Low Literacy | 1 | 3 | 4
    Marginal Literacy | 28 | 29 | 57
    Adequate Literacy | 165 | 159 | 324

OUTCOME MEASURES:

1. Primary Outcome: Planning Behavior Score at 1-month
Description: The primary endpoint for this study is planning behavior score (ranging from 5-25 points; where higher values are considered to be a better outcome) at one month post-intervention/attention control as measured by the "Planning Implementation (Behavior)" assessment. The outcome measure will be assessed at baseline and one month from baseline. Primary endpoint analyses will consist of an analysis of covariance (ANCOVA) comparing mean planning behavior score at one month post-intervention/attention control while controlling for baseline planning behavior score. All analyses will assume a type I error rate of 5%.
Time Frame: baseline and 1 month
Population: All randomized participants with a complete planning behavior score at baseline and one-month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plan Your Lifespan Website | Go4Life Website
Number analyzed (Participants) | 167 | 179
units on a scale
  Baseline Planning Behavior Score | 16.97 (4.38) | 16.80 (4.58)
  One Month Planning Behavior Score | 17.19 (4.48) | 15.88 (4.56)
Statistical Analysis 1: Comparison: Plan Your Lifespan Website vs Go4Life Website; H1: Compared to participants in the attention control group and controlling for baseline assessments, participants receiving the PLAN YOUR LIFESPAN tool will show increased planning with regard to planning behavior score (measured via the Planning Assessment tool) one (efficacy) month after intervention; Test type: Superiority or Other; p = 0.0054, ANCOVA; Slope = 1.25, 95% CI 2-sided [0.37 to 2.12], Standard Error of Mean 0.45

2. Secondary Outcome: Planning Perception Score at Baseline, Immediate Post-test, 1 and 3-months
Description: Planning perception score (ranging from 5-25 points where higher values are considered to be a better outcome) at all follow-up time points as measured by the "Planning Perception" assessment. This secondary outcome measure will be assessed at baseline, immediate post-test, 1, and 3-months.
Time Frame: baseline, post-intervention, 1 month, and 3 months
Population: Participants with a complete baseline planning behavior score and either a complete one-month or three-month planning behavior score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plan Your Lifespan Website | Go4Life Website
Number analyzed (Participants) | 179 | 183
units on a scale
  Baseline Planning Perception Score | 19.75 (4.02) | 20.11 (3.64)
  Post-Tool Planning Perception Score | 20.70 (3.85) | 20.01 (3.74)
  One-Month Planning Perception Score | 20.75 (3.69) | 20.29 (3.61)
  Three-Month Planning Perception Score | 21.14 (3.55) | 20.81 (3.56)
Statistical Analysis 1: Comparison: Plan Your Lifespan Website vs Go4Life Website; Secondary analyses will compare baseline variables (current utilization of services, physical function assessment, co-morbidities, social support, health literacy, self-efficacy, and sociodemographics) with outcome (one-at-a-time). Those found to have a significant association with outcome will be included in a linear mixed model, with random effect for intercept. A backward stepwise model building process will be used to determine an overall parsimonious model for outcome; Test type: Superiority or Other; p = 0.0471, Mixed Models Analysis — P-value controlled for significant baseline covariates (sex, importance of religion, stroke, and self efficacy score) and individual participant effect; The p-value is based on the slope estimation provided below; Slope = 0.244, Standard Error of Mean 0.123

3. Secondary Outcome: Confidence in Accessing Home Services Score at Immediate Post-test, 1 and 3-months
Description: Participant confidence in accessing home services based on a 5-item questionnaire. The score is the equally-weighted sum of responses to the five questions in the CAHS instrument. Each question has a scale of 1-5, giving a total possible range of 5-25, with 5 representing low confidence and 25 representing high confidence. No subscores are calculated.
Time Frame: baseline, post-intervention, 1 month, and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plan Your Lifespan Website | Go4Life Website
Number analyzed (Participants) | 179 | 183
units on a scale
  Baseline CAHS Score | 20.85 (3.29) | 20.70 (3.45)
  Post-Tool CAHS Score | 21.39 (2.89) | 20.67 (3.37)
  One-Month CAHS Score | 21.74 (2.62) | 21.19 (2.93)
  Three-Month CAHS Score | 22.17 (2.33) | 21.70 (2.71)
Statistical Analysis 1: Comparison: Plan Your Lifespan Website vs Go4Life Website; H2: Compared to participants in the attention control group and controlling for baseline assessments, participants receiving the PLAN YOUR LIFESPAN tool will show increased confidence in accessing home services (measured via the Confidence in Accessing Home Services tool) one (efficacy) and three (effect retention) months after intervention; Test type: Superiority or Other; p = 0.423, Mixed Models Analysis — p-value controlled for significant baseline covariates (confidence in using the internet, self efficacy score, support score, and race/ethnicity; The p-value is based on the slope estimation provided below; Slope = 0.075, Standard Error of Mean 0.094 — The score is the equally-weighted sum of responses to the five questions in the CAHS instrument. Each question has a scale of 1-5, with a total possible range of 5-25. No subscores are calculated

4. Secondary Outcome: Knowledge of Home Services Score at Immediate Post-test, 1 and 3-months
Description: Knowledge of home services score at all follow-up time points as measured by "Understanding of Home Services" assessment. This is a 6-item knowledge assessment; each question is scored as correct or incorrect and questions are equally weighted. The total possible range of scores is 0-6,with 0 being low knowledge and 6 being high.
Time Frame: baseline, post-intervention, 1 month, and 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Plan Your Lifespan Website | Go4Life Website
Number analyzed (Participants) | 179 | 183
units on a scale
  Baseline UHS Score | 3.56 (1.28) | 3.79 (1.27)
  Post-Tool UHS Score | 4.12 (1.26) | 3.93 (1.21)
  One-Month UHS Score | 4.10 (1.35) | 3.72 (1.39)
  Three-Month UHS Score | 4.18 (1.45) | 3.73 (1.37)
Statistical Analysis 1: Comparison: Plan Your Lifespan Website vs Go4Life Website; Compared to participants in the attention control group, participants receiving PLAN YOUR LIFESPAN will show increased UHS 1 (efficacy) and 3 (effect retention) months post-intervention. Secondary analyses will compare baseline variables with outcome (one-at-a-time). Those with a significant association with outcome will be included in a LMM for UHS, with random effect for intercept. A backward stepwise model building process will be used to determine an overall parsimonious model for UHS; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value controlled for significant baseline covariates (sex, income, health literacy, education level, high blood pressure, and kidney disease) and individual participant effect; The p-value is based on the slope estimation provided below; Slope = 0.22, Standard Error of Mean 0.05

5. Secondary Outcome: Satisfaction With Intervention Tool Score at Immediate Post-test, 1 and 3-months
Description: Overall satisfaction with the intervention or attention control as measured by the "Satisfaction with Intervention Tool." Tests will be performed at a two-sided 5% significance level.
Time Frame: baseline, post-intervention, 1 month, and 3 months
Population: Due to errors in the data collection method, it is not possible to summarize the data for reporting.
Groups:
- Plan Your Lifespan Website: Participants in the intervention arm will navigate the Plan Your Lifespan website, a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas described below.
  Plan Your Lifespan Website: Participants in the intervention arm will navigate the advance planning tool, Plan Your Lifespan, a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. A minimum of 15 minutes and a maximum of 45 minutes will be allotted for navigating this website.The Plan Your Lifespan website is also interactive in that it allows participants to enter their information and share it with others to facilitate conversations and decision-making.
Arm/Group | Plan Your Lifespan Website | Go4Life Website
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Plan Your Lifespan Website: Participants in the intervention arm will navigate PlanYourLifespan.org, a Web-based planning tool that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. PlanYourLifespan.org is also interactive in that it allows participants to enter their information and share it with others to facilitate conversations and decision-making.
  PlanYourLifespan.org: Participants in the intervention arm will navigate PlanYourLifespan.org, that provides information for seniors related to advanced health planning for home services in specific content areas of: hospitalizations, falls, Alzheimer's, dementia, as well as communicating with others. A minimum of 15 minutes and a maximum of 45 minutes will be allotted for navigating this website.
Arm/Group | Plan Your Lifespan Website | Go4Life Website
Serious Adverse Events (participants affected / at risk) | 0/194 | 0/191
Other Adverse Events (participants affected / at risk) | 0/194 | 0/191

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No